CLINICAL TRIAL: NCT04352933
Title: ChemoPROphyLaxIs For covId-19 Infectious Disease (the PROLIFIC Trial)
Brief Title: PROLIFIC ChemoprophylaxisTrial (COVID-19)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Joseph Cheriyan, MD, Dr, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PROLIFIC2020 (A095583)
Record Dates: First submitted 2020-04-07; First posted 2020-04-20 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Coronavirus; COVID-19; chemoprophylaxis; Hydroxychloroquine
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydroxychloroquine - Daily dosing (Active Comparator): Hydroxychloroquine Daily (loading phase: 800mg for first 2 days; maintenance phase: 1 x 200mg tablet every day) + weekly placebo, for approximately 90 days.
  Route: Oral. Pharmaceutical form: Tablet
  Interventions: Drug: Hydroxychloroquine - Daily dosing
- Hydroxychloroquine - Weekly dosing (Active Comparator): Hydroxychloroquine weekly (loading phase: 800mg for first 2 days; maintenance phase: 2 x 200mg tablets every 7th day/weekly) + daily placebo, for approximately 90 days.
  Route: Oral. Pharmaceutical form: Tablet
  Interventions: Drug: Hydroxychloroquine - Weekly Dosing
- Placebo (Placebo Comparator): Placebo arm - 2 tablets twice daily for first 2 days (loading phase), followed by 1 tablet every day for 90 days plus 2 tablets every 7th day, for approximately 90 days.
  Route: Oral. Pharmaceutical form: Tablet
  Interventions: Other: Matched Placebo Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine - Daily dosing — Active HCQ:
  Days 1-2: Loading phase - 400mg (2 x 200mg capsules) taken TWICE A DAY for 2 days Days 3 onwards: Maintenance Phase - 200mg (1 x 200mg capsule) taken ONCE A DAY, every day for 90 days (~3 months),
  Matched Placebo HCQ:
  Days 3 onwards: Maintenance Phase - 2 capsules taken ONCE A WEEK on the same day each week (every 7th day) for 90 days (~3 months)
  Arms: Hydroxychloroquine - Daily dosing
Drug: Hydroxychloroquine - Weekly Dosing — Active HCQ:
  Days 1-2: Loading Phase - 400mg (2 x 200mg capsules) taken TWICE A DAY for 2 days Days 3 onwards: Maintenance Phase - 400mg (2 x 200mg capsules) taken ONCE A WEEK on the same day each week (every 7th day) for 90 days (~3 months)
  Matched Placebo HCQ:
  Days 3 onwards: Maintenance Phase - 1 capsule taken ONCE A DAY for 90 days (~3 months)
  Arms: Hydroxychloroquine - Weekly dosing
Other: Matched Placebo Hydroxychloroquine — Matched placebo HCQ - daily dosing:
  Days 1-2: Loading Phase - 2 capsules taken TWICE A DAY for 2 days Days 3 onwards: Maintenance Phase - 1 capsule taken ONCE A DAY for 90 days (~3 months) Matched placebo HCQ - weekly dosing Days 3 onwards: Maintenance Phase - 2 capsules taken ONCE A WEEK on the same day each week (every 7th day) for 90 days (~3 months)
  Arms: Placebo

SUMMARY:
The number of confirmed cases of COVID-19 infectious disease arising from the SARS-CoV-2 coronavirus is rising substantially and rapidly, with the potential to overwhelm the ability of the entire National Health Service (NHS) to cope with the increased demand. The availability of personal protective equipment is limited and reports of high risk procedures such as aerosol generating procedures (e.g. intubation for the sickest patients) is a source of great concern for infection transmission. Frontline NHS staff with direct patient contact have the highest likelihood of exposure to SARS-CoV-2 and development of COVID-19 disease. Efforts to protect these workers from development of COVID-19, using drugs to prevent the disease, require urgent evaluation.

DETAILED DESCRIPTION:
The number of confirmed cases of COVID-19 infectious disease arising from the SARS-CoV-2 coronavirus is rising substantially and rapidly, with the potential to overwhelm the ability of the entire National Health Service (NHS) to cope with the increased demand. The availability of personal protective equipment is limited and reports of high risk procedures such as aerosol generating procedures (e.g. intubation for the sickest patients) is a source of great concern for infection transmission. Frontline NHS staff with direct patient contact have the highest likelihood of exposure to SARS-CoV-2 and development of COVID-19 disease. Efforts to protect these workers from development of COVID-19, using drugs to prevent the disease, require urgent evaluation.

This trial will be a double-blind, randomized, placebo-controlled trial in a cohort of frontline healthcare workers, who will potentially be exposed to SARS-CoV-2. Eligible participants will be frontline NHS workers aged 18 to 70 years who work in a healthcare setting with direct patient care. Participants will be randomised to one of 3 arms and receive either: (1) Hydroxychloroquine Daily (loading phase: 800mg for first 2 days; maintenance phase: 1 x 200mg tablet every day) + weekly placebo; (2) Hydroxychloroquine weekly (loading phase: 800mg for first 2 days; maintenance phase: 2 x 200mg tablets every 7th day/weekly) + daily placebo, or (3) placebo (daily and weekly).

Participants will be reviewed at an interim visit 6 weeks after baseline and again and the end of the study treatment in 90 days (approximately 3 months) after randomization. Participants will also complete brief questions about their health weekly while on treatment (remotely, via app/web/phone-based interface).

ELIGIBILITY:
Inclusion Criteria:

To be included in the trial the participant MUST:

1. Have given written informed consent to participate
2. Be aged 18 years to 70 years
3. Not previously have been diagnosed with COVID-19
4. Work in a high-risk secondary or tertiary healthcare setting (hospitals accepting COVID-19 patients) with direct patient-facing care

Exclusion Criteria:The presence of any of the following will mean participants are ineligible:

1. Known COVID-19 positive test at baseline (if available)
2. Symptomatic for possible COVID-19 at baseline
3. Known hypersensitivity reaction to HCQ, chloroquine or 4-aminoquinolines
4. Known retinal disease
5. Known porphyria
6. Known chronic kidney disease (CKD; eGFR<30ml/min)
7. Known epilepsy
8. Known heart failure or conduction problems
9. Known significant liver disease (Gilbert's syndrome is permitted)
10. Known glucose-6-phosphate dehydrogenase (G6PD) deficiency
11. Currently taking any of the following contraindicated medications:

    1. Digoxin
    2. Chloroquine
    3. Halofantrine
    4. Amiodarone
    5. Moxifloxacin
    6. Cyclosporin
    7. Mefloquine
    8. Praziquantel
    9. Ciprofloxacin
    10. Clarithromycin
    11. Prochlorperazine
    12. Fluconazole
12. Currently taking hydroxychloroquine or having a clinical indication for taking hydroxychloroquine
13. Currently breastfeeding
14. Unable to be followed-up during the trial
15. Current or future involvement in the active treatment phase of other interventional research studies (excluding observational/non-interventional studies) before study follow-up visit
16. Not able to use or have access to a modern phone device/web-based technology
17. Any other clinical reason which may preclude entry in the opinion of the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Time to positive COVID-19 disease | Assessed up to 90 days
  Time taken for incidence of COVID-19 disease between Hydroxychloroquine and placebo arms

SECONDARY OUTCOMES:
Number of COVID-19 test positive cases | Assessed up to 90 days
  Number of COVID-19 symptoms based on clinical guidelines and test positive infections per study arm
Number of COVID-19 serological test positive cases | Assessed up to 90 days
  Number of test positive COVID-19 serological test positive cases per study arm
Severity of COVID-19 disease between each arm | Assessed up to 90 days
  Severity based on hospitalisation
Number of common COVID-19 complications between each arm | Assessed up to 90 days
  Number of common COVID-19 complications between arms

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cheriyan, MBCHB, FRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No